CLINICAL TRIAL: NCT07053787
Title: Durability of Yoga for Treating Veterans With Chronic Low Back Pain
Brief Title: Durability of Yoga for Veterans With Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRD2-001-24W
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; yoga; disability; durability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The trial is a single blind RCT as participants will be exposed to the study conditions allocated but will be unaware of the study hypotheses and details of the differences between the two yoga conditions. At follow-up assessments, assessors will be blinded to the participant group assignment and participants will be asked not to discuss their group assignment when contacted by staff. The investigators will be blinded to group assignment. Only the Study Coordinator is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Yoga (Active Comparator): Hatha yoga designed for Veterans with chronic low back pain.
  Interventions: Behavioral: Standard Yoga
- Enhanced Yoga (Experimental): Hatha yoga designed for Veterans with chronic low back pain plus coaching and texts to enhance durability and long-term adherence to yoga.
  Interventions: Behavioral: Enhanced Yoga

INTERVENTIONS:
Behavioral: Standard Yoga — Weekly hatha yoga for 12 weeks augmented by home practice guided by yoga instructional videos.
  Arms: Standard Yoga
Behavioral: Enhanced Yoga — Weekly hatha yoga for 12 weeks augmented by home practice guided by yoga instructional videos ...
  plus six weekly 50-minute 1-on-1 coaching sessions starting week 10 of the standard yoga intervention and ending week 15 (3 wks after end of standard yoga). During this transition, participants are supported with development and execution of their plan for continuing their yoga practice. Participants will be offered 1 additional ad-hoc coaching session to help them re-start yoga if they get off track and/or experience major life events such as moving, job change, medical issues, etc.
  Arms: Enhanced Yoga

SUMMARY:
Chronic low back pain is a prevalent condition among VA patients, but many current treatment options have side effects or limited effectiveness. Veterans with chronic low back pain (cLBP) experience increased disability, functional challenges, and reduced quality of life. A prior VA funded study of Yoga for VA patients with cLBP found that yoga can reduce pain and disability at 3 and 6 months after enrollment. However, the long-term effects and maintenance of yoga practice is unknown. The current study will test an intervention designed to promote long-term yoga practice and long-term health outcome benefits at 12 and 18 months after enrollment.

DETAILED DESCRIPTION:
Significance to VA:

Chronic low back pain (cLBP) is a highly prevalent condition for veterans. In addition to chronic pain, cLBP leads to significant amounts of disability, reduced health-related quality of life (QOL), and increased health care utilization. Our previous results and other studies of yoga for Veterans with cLBP show that yoga participants had reduced pain and disability at follow-up assessments at 6-month follow-up. There is also some evidence indicating that self-care treatments like yoga, especially those provided in group format, may be less expensive and may reduce health care costs, conserving limited resources for other conditions and services. Since persons with cLBP usually live with this chronic condition for the rest of their lives, understanding and facilitating long-term yoga practice for VA patients is an important step for the provision of high-quality VA healthcare.

Innovation and Impact:

If funded, this will be the first study to examine a durability intervention for promoting long-term yoga practice. It uses text messaging for both behavioral reminders, and for ecological momentary assessment of the durability outcome. The study tracks 18 months of follow-up data.

Specific Aims:

The primary aims of the proposed project are to examine the effectiveness of a coaching intervention plus text reminders for promoting long-term maintenance of yoga practice and function among Veterans with cLBP. The investigators will also examine intervention costs and subsequent health care costs.

Methodology:

The investigators will recruit and randomize 176 Veterans with cLBP to either standard yoga or the durability-enhanced yoga intervention. Participants will complete health outcome assessments at baseline, 3 months, 6 months, 12 months, and 18 months. The standard yoga intervention includes weekly in-person yoga sessions for 12 weeks. The enhanced yoga arm will receive weekly behavioral coaching sessions from weeks 10-15 and will receive ongoing text reminders. The co-primary outcomes will be the mean days and minutes per week of yoga practice and the mean change in back pain-related disability at 12 months. The investigators will measure yoga practice and other health outcomes including pain severity, QOL, and fatigue through 18 months. The investigators will measure attendance and home practice. The investigators will monitor and assess adverse events and instructor fidelity.

Path to Translation/Implementation:

If the durability intervention can increase long-term yoga practice and associated health benefits, this will provide very strong evidence for wider implementation of yoga as a specific treatment for chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* VA patients > 18 years
* Diagnosis of chronic low back pain > 3 mos
* Pain rated 4/10 or higher
* No new pain treatments in the past month.
* Willing to attend intervention;
* Complete 5 assessments;
* Respond to text assessments
* Practiced yoga < 3x in the last 6 months
* Unless medically necessary, agree to not change pain treatment during intervention

Exclusion Criteria:

* Back surgery within the last 1 year
* Pain due to specific systemic (eg, scleroderma, fibryomalgia) or non-musculoskeletal problem (neuropathy)
* Positive Romberg test (with or without sensory neuropathy)
* Severe vertebral disk problems, sciatica or nerve compression >3 months
* Serious or unstable psychiatric illness (e.g., unmanaged psychosis, manic episode, or substance dependence)
* Serious coexisting medical illness (eg, cancer, COPD, bmi> 40)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Days and minutes per week of yoga practice - Ecological Momentary Assessment (EMA) of Yoga | Baseline to 18 months
  The investigators will employ EMA to assess weekly yoga practices across the whole 18-month study period. Because yoga includes both mind and body components, as well as movements that are not aerobic in nature, yoga cannot be assessed like other physical activities using accelerometers. EMA has been shown to enhance self-report because it occurs randomly, so as not subject to recall bias, and frequently so is not subject to recall errors. The investigators will ask how many minutes of yoga, if any, have been performed on the assessment day and whether it was performed at home or at an in-person class. Participants will receive an EMAs every week across the 18-monthstudy period. If participants do not respond within 90 minutes, a reminder will be sent. If there is still no response, they will be sampled again in the next 24 hours at a different time of day.
Roland-Morris Disability Questionnaire | Change from baseline to 18 months
  The RMDQ will serve as the primary health outcome and consists of 23 questions about limitations experienced for a variety of daily activities. The scale has been shown to be reliable and is well validated. It has been used in other studies of yoga studies. Scores range from 0 to 23, with higher scores indicating more back pain-related disability.

SECONDARY OUTCOMES:
Pain Severity - Brief Pain Inventory (BPI) | Change from baseline to 18 months
  This subscale assesses pain severity using a Numeric Rating Scale (NRS) from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable. The mean of multiple items is used. Higher mean scores indicate greater pain severity.
Pain Interfernce - Brief Pain Inventory (BPI) | Change from baseline to 18 months
  This subscale assesses pain interference using a Numeric Rating Scale (NRS) from 0 to 10, where 0 is no pain and 10 is the worst pain interference imaginable. The mean of multiple items is used. Higher mean scores indicate greater pain interference.
Fatigue - Fatigue Severity Scale (FSS) | Change from baseline to 18 months
  The Fatigue Severity Scale (FSS) has a score range of 9 to 63. Higher scores indicates more severe fatigue.
Quality of Life - SF12 | Change from baseline to 18 months
  Physical and mental QOL will be assessed with the Short-form 12 (SF12). The SF-12 uses a norm-based scoring system, where the mean score for the general population is 50, and standard deviation is 10. Scores range from 0 to 100, with higher scores indicating better QOL/ health status.
Yoga Self-Efficacy Scale (YSES) | Change from baseline to 18 months
  YSES scores range from 12 to 108, with higher scores indicating greater perceived self-efficacy in yoga practice.

OTHER OUTCOMES:
Health Care utilization and costs | Baseline to 18 months
  Health care utilization data for participants will be obtained from the VA Corporate Data Warehouse (CDW). Utilization data are converted to estimated costs using costing algorithms from VA HERC. Costs are stated in US$.

CONTACTS AND LOCATIONS:
Overall Officials: Erik J. Groessl, PhD BA BS, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared.
Supporting Information: Study Protocol
Time Frame: 12 months after study completion to allow for results to be published. Data will be available indefinitely.
Access Criteria: Requests for access to this data must be made in writing signed by a requestor from the United States. The request should reference the publication underlying the request. Requests may be made to the Principal Investigator/lead point-of-contact for the publication. Should the investigator leave the VASDHS, the requests may be sent to the Associate Chief of Staff for Research.